CLINICAL TRIAL: NCT00050843
Title: A Study to Access the Safety/Efficacy of Thalidomide in the Treatment of Anemia in Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: Celgene (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THAL-MDS-001
Record Dates: First submitted 2002-12-23; First posted 2002-12-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-05

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
The primary objective of the study is to determine the efficacy of thalidomide for the treatment of anemia in patients with myelodysplastic syndromes (MDS).

ELIGIBILITY:
* Eligible patients must have a diagnosis of myelodysplastic syndrome
* Life expectancy of at least 6 months.
* Patients must be able to adhere to the study visit schedule and other protocol requirements.
* Patients must understand and voluntarily sign an informed consent document.
* Women of childbearing potential (WCBP) must agree to practice abstinence or to use TWO methods of contraception beginning 4 weeks prior to the start of study medication and throughout the course of treatment.
* Males must use barrier contraception when engaging in reproductive sexual activity with women of childbearing potential.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2001-08; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Scripps Cancer Center, La Jolla, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Desert Hematology Oncology Medical Group INC, Rancho Mirage, California
  - Whittingham Cancer Center, Norwalk, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Southeast Florida Hematology-Oncology, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northwest Medical Specialists, Arlington Heights, Illinois
  - Oncology Associates, Cedar Rapids, Iowa
  - Beaumont Cancer Center, Royal Oak, Michigan
  - SMDC Health Systems, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Jackson Oncology Associates PLLC, Jackson, Mississippi
  - Hematology Oncology Consultants Inc, St Louis, Missouri
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hematology Oncology Associates of NJ, Paramus, New Jersey
  - Summit Medical Group/Overlook Oncology Center, Summit, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - VAMC Northport, Northport, New York
  - University of Rochester Cancer Center, Rochester, New York
  - South Shore Hem-Onc Assoc. PA, Rockville Centre, New York
  - Staten Island Unversity Hospital, Staten Island, New York
  - Westchester County Medical Center, Valhalla, New York
  - Buffalo Medical Group PC, Williamsville, New York
  - Northwestern Carolina Hematology Oncology PA, Hickory, North Carolina
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Oncology/Hematology Care Inc, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Lancaster Cancer Center LTD, Lancaster, Pennsylvania
  - MCP Hahnemann University, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Texas Oncology PA-BMT Center, Dallas, Texas
  - Central Utah Medical Clinic, Provo, Utah
  - InterMountain Hematology/Oncology, Salt Lake City, Utah
  - Swedish Cancer Institute, Seattle, Washington
  - Yakima Regional CancerCenter, Yakima, Washington